CLINICAL TRIAL: NCT06047925
Title: 3D-printed Crowns Versus Prefabricated Stainless-Steel Crowns for Intermediate Restoration of Compromised First Permanent Molars (Randomized Controlled Clinical Trial)
Brief Title: 3D-printed Crowns Versus Prefabricated Stainless-Steel Crowns for Intermediate Restoration of Compromised First Permanent Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Bassam Mohamed Ahmed, Asisstant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-RECID022321
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: 3D Printed Crowns
Keywords: 3D printed crowns- Stainless steel crowns

STUDY DESIGN:
Intervention Model Description: one experimental group and one active comparator group
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator-outcome Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): First permanant molar will be prepared to receive 3D printed crown
  Interventions: Procedure: 3D printed crown
- group B (Active Comparator): First permanant molar will be prepared to receive SSC
  Interventions: Procedure: stanless steel crown

INTERVENTIONS:
Procedure: 3D printed crown — Reduction will be performed on the occlusal surface using a flame stone or a wheel stone, to perform occlusal clearance by 1 mm. Reduction will be performed by 1 mm on the mesial, distal, buccal and lingual surfaces of the tooth. Impression for the preparation will be taken using putty and light poly vinyl siloxane material. Temporary crown will be placed above the preparation as temporisation.The impression will be sent to the lab .The preparation will be optically scanned in the lab and the restoration will be digitally designed using computer designing software.The crown will be printed using 3D printer using hybrid resin(micro-filled hybrid material) material.The 3d printed crown is cemented with resin cement.
  Arms: group A
Procedure: stanless steel crown — The occlusal surface of the tooth should be reduced by about 1.5 mm, maintaining its occlusal contour or until the tooth is out of occlusion with adequate room to fit a crown.Proximally, tooth reduction will be made through the mesial and distal contact areas, then roundation of line angles to avoid the creation of ledges or steps.The crown selection will be done by trial and error or by measuring the mesiodistal dimension of the tooth space with dividers. It can also be helpful to measure the dimension of the contralateral tooth. A correctly fitting crown should snap or click at try in.
  Arms: group B

SUMMARY:
The study will evaluate the clinical performance and both patient and parent satisfaction of 3d printed crowns versus prefabricated Stainless-steel crowns (SSCs) in compromised first permanent molars

DETAILED DESCRIPTION:
A total of Forty permanent first mandibular molars in healthy subjects will be selected from the Pediatric Dentistry and Dental Public Health outpatient clinic.

The molars will be randomly assigned equally into two treatment groups group A 3D-printed crowns & group B prefabricated SSCs, removal of caries with a high-speed handpiece then removal of the remaining carious lesion with excavator then glass ionomer restoration will be placed, preparation of SSCs crowns will be done in Group A by reduction of occlusal surface by about 1.5 mm, Proximally, tooth reduction is made through the mesial and distal contact areas, then roundation of line angles. Proper size of crown will be selected. It can also be helpful to measure the dimension of the contralateral tooth. A correctly fitting crown should snap or click at try in. In group B reduction will be performed on the occlusal surface using a flame stone or a wheel stone, to perform occlusal clearance. Reduction will be performed on the mesial, distal, buccal, and lingual surfaces of the tooth Then roundation of the line angles will be performed. Impression for the preparation will be taken using putty and light poly vinyl siloxane material. The preparation will be optically scanned in the lab and the restoration will be digitally designed using computer designing software. The crown will be printed using 3D printer using hybrid resin material. Crown will be checked for proper fit and cemented to the tooth by self-etch adhesive.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the study should conform to the following criteria:

  1. Badly broken-down endodontically treated first permanent molar
  2. First permanent molar with extensive multi-surface caries.
  3. First permanent molar with structural developmental defects such as hypoplasia, Molar-Incisor Hypomineralization (MIH), Amelogenesis Imperfecta, and Dentinogenesis Imperfecta

Exclusion Criteria:

* Children who are uncooperative needing sedation or general anesthesia.
* Children who are physically or mentally disabled or having any medical condition that will complicate the treatment.
* Molars of poor prognosis

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The clinical performance of 3d printed crowns versus prefabricated SSCs in compromised first permanent molars | 3,6,12 and 18 months
  Evaluation of clinical performance of both crowns regarding gingival health (gingival & plaque index) and Fracture, retention, marginal discoloration and surface texture according to the modified United states Public Health Service (USPHS) criteria. 3,6-12 and 18 months.

SECONDARY OUTCOMES:
Patient and parent satisfaction. | Immediately ,3,6,12&18 months
  Parental and patient satisfaction will be assessed during the delivery session to determine their satisfaction level with 5-point Likert scale where 1-very dissatisfied; 2-dissatisfied; 3-neutrally satisfied; 4-satisfied; 5-very satisfied. Child's perception regarding their esthetics with crowns will be also considered in this study. Children will be asked to rank the crowns based on "Smiley Face Likert Scale."

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa khattab, BDS,MSc,MD, Study Director — Ainshams University
Locations (1):
- Faculty of dentistry Ainshams university, Cairo, Egypt